CLINICAL TRIAL: NCT05742815
Title: Nationwide Sampling of Donor Human Milk Nutrient Content
Brief Title: Analysis of Donor Milk
Acronym: DOME
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Amy Gates, Adjunct Intructor, Augusta University
Other Study IDs: 1823198-1
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Breast Milk Collection; Nutrition Disorder, Infant
MeSH Terms: conditions — Breast Milk Expression; Infant Nutrition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational collection of data from purchased donor milk samples

SUMMARY:
The purpose of this prospective, cross-sectional, observational study is to measure the nutrient composition of donated human breastmilk purchased from commercial human milk banks in North America

DETAILED DESCRIPTION:
Aim 1: To measure the micronutrient, macronutrients, microbial count, and endotoxins present in donated human breastmilk purchased from commercial human milk banks in North America (Table 2).

Aim 2: To compare the results of the nutrient analysis to nutrient recommendations for premature infants. (Table 3).

Aim 3: To use the results of the nutrient analysis to calculate the final nutrient content of donor human milk after the addition of commonly used human milk fortifiers (HMF). We will compare the calculated nutrients with intake recommendations for premature infants.

Background Preterm infants are at risk for nutrition depletion because of inadequate placental transfer, low volume feedings in the first days of life, and increased nutrient needs.1-3 Adequate intake of nutrients during neonatal development is crucial for growth. In addition, preterm infants are vulnerable to feeding-related complications, including necrotizing enterocolitis (NEC) and enteral feeding intolerance.4,5 Human milk feedings reduce the risk of NEC and enteral feeding intolerance and are considered the standard of feeding for this population. When mother's own milk (MOM) is not available or is inadequate to meet the needs of the infant, donor human milk (DHM) is the recommended feeding choice for preterm infants with birth weights ≤1500 grams.5 Several factors influence the nutrient composition of human milk, including lactation stage, gestational age at delivery, maternal age, body mass index (BMI), diet, and race.6-8 Preterm MOM is more nutrient-dense than mature human milk and continues to change as the lactation stage progresses.6,7,9 Donors of human milk are typically mothers of infants born at term and are unlikely to donate milk in the first month after delivery when milk is most nutrient-dense.

In 2011 22% of American neonatal intensive care units (NICU) used DHM to feed preterm infants. By 2017 the number of NICU purchasing DHM increased to 75%.10 To meet the demand for DHM, the number of human milk banks has increased from two in 1985 to more than thirty in 2020. The human milk banking industry is self-regulated with little oversight from governmental agencies. Donor human milk can be purchased from non-for-profit, private, public-benefits companies, or mother's milk co-operatives. Practices for donor selection, milk pooling, pasteurization or sterilization, nutrient analysis, and labeling vary by bank.11 Most DHM banks in North America do not report the nutrient composition of the DHM they sell. Of those that do, only three report nutrients other than protein, energy, and fat. Understanding the nutrient profiles of DHM is essential for creating feeding plans to meet the needs of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Donor human milk from commercially available milk banks

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Donor milk samples will be collected from commercially available donor milk banks
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Nutrient composition of donor human milk samples | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gates A, Maria SD, Meredith NA, Houslay T, Stansfield BK. Vitamin A in donor human milk: An experimental study. JPEN J Parenter Enteral Nutr. 2025 Nov;49(8):951-954. doi: 10.1002/jpen.70008. Epub 2025 Aug 20. PMID 40836482
- [Derived] Gates A, Hair AB, Salas AA, Thompson AB, Stansfield BK. Nutrient Composition of Donor Human Milk and Comparisons to Preterm Human Milk. J Nutr. 2023 Sep;153(9):2622-2630. doi: 10.1016/j.tjnut.2023.07.012. Epub 2023 Jul 28. PMID 37517552